CLINICAL TRIAL: NCT04287764
Title: Repeatability of the Infant Food Reinforcement Paradigm: Implications of Individual and Developmental Differences
Brief Title: Infant Test-Retest of the Food Reinforcing Ratio Task
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Collaborators: research institute on addictions (Unknown)
Responsible Party: Principal Investigator, Kai Ling Kong, Principal Investigator, State University of New York at Buffalo
Other Study IDs: Test Re-test
Record Dates: First submitted 2020-02-24; First posted 2020-02-27 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Infant Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess the test-retest reliability of an infant RRV paradigm which will allow researchers to study food reinforcement among infant of 9-18 months of age. By understanding the origins of food reinforcement, future interventions can be conducted to help overweight and obese population to alter their reinforcing values of food at a young age, perhaps during infancy.

DETAILED DESCRIPTION:
1. Initial email or phone screen:

   Upon receiving an inquiry from a prospective participant, the study will be explained. If the prospective participant has an infant age 9 to 18 months, and the caregiver is interested in joining the study, a verbal consent will be obtained in order to screen for eligibility criteria. The initial screening questionnaire could be done via phone or online via Survey Monkey (see Initial Phone Screen/Survey Monkey Questionnaire for details). The information assessed during the initial screen is recorded in a secure database that requires a password. The database is used by select members of the Division of Behavioral Medicine and has been approved for use by previous IRB committees.

   Families will also be sent a list of links of questionnaires to be completed at home before the assessments. These questionnaires include the Demographic Questionnaire, Pregnancy History and Infant Feeding Practice Questionnaire, Food Security Questionnaire, Infant Behavior Questionnaires-Revised (IBQ-R), and Baby Eating Behavior Questionnaire (BEBQ).
2. Session 1:

   If families meet the initial criteria gathered from the initial screen, families will be scheduled for a laboratory visit (40 min). For this visit, the caregiver will be advised to choose a time of the day when the infant is generally alert, active, and ready to play. The infant needs to be fed one hour prior to the lab visit. The caregiver will be reminded to bring diapers or change of clothes for the infant. The caregiver will also be reminded not to feed her infant the test food (infant's favorite food) 24 hours before the laboratory visit. At the first visit, there will be an overview of the study. If interested, the caregiver will be asked to review and sign consent forms. Two copies of the consent forms will be signed by all parties involved, person obtaining consent, and the participating parent. One copy will be obtained by the study personnel and one copy will be given to the participants for their records. The copy obtained by study personnel will be kept in a locked cabinet.

   After signing the consent form, the caregiver and infant will be escorted to a laboratory room where the food reinforcement game will take place. At this visit, infant will play the first part of the RRV game. Infants will be securely fastened on a high chair. The caregiver will be in the room with the infant at all-time during the game. The caregiver will be reminded that the entire reinforcement task procedure will be video recorded to obtain vocalization, body movement, and facial expression of the infant. The baseline state of the infant will be assessed. There are five states: 1 = drowsy, 2 = alert/calm, 3 = alert/active, 4 = fussy, 5 = crying. Before the start of the game, a study staff member will go through a training session with the infant to familiarize him/her with the computer based game and button/monitor interface. The caregiver will be asked to assist with the training by repeating phrases the researchers use during the game. After the training, the study staff member will start the actual game.

   After the session is finished, a 3-day dietary recall will be conducted via phone by a dietetic student intern
3. Additional Laboratory Sessions:

Participants are invited to attend 3 additional 40 minute laboratory sessions. For these visits, the infants will be playing the second part of the RRV game (please refer Session 1 for details on the game), and then repeat RRV Games parts 1 and 2 on the subsequent laboratory visits. After Sessions 1, 2, and 3, the dietetic student intern will call the caregiver and conduct a 24-hour dietary recall. Before leaving the last visit, the height and weight of the caregiver and infant will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Infant must be between the ages of 9 to 18 months old
* Infant must appear to be healthy
* Infant of singleton (i.e. not twin or multiple)
* Infant not allergic to puffed grains or Original Cheerios

Exclusion Criteria:

* Infant of pre-mature or pre-term birth (< 37 weeks of gestation)
* Infant of low birth weight (<2500 grams)
* Infant with medical problems at birth
* Infant with developmental delay based on developmental milestones recorded at 6 or 9 month check up
* Infant who has not eaten the test food due to allergy concern
* Maternal age < 18 years
* Mother who smoked, used controlled substances (i.e. opiates, cocaine, marijuana) or consumed excessive alcohol during pregnancy
* Mother who had a high-risk pregnancy

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants ages 9-18 months
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
FRR | through study completion, an average of 1 year
  The primary outcome is the reliability of the food reinforcing ratio.

SECONDARY OUTCOMES:
Weight status | through study completion, an average of 1 year
  The secondary outcome measures are infant weight status

CONTACTS AND LOCATIONS:
Overall Officials: Kai ling Kong, Principal Investigator — Assistant Professor